CLINICAL TRIAL: NCT07358312
Title: Traumatic Brain Injury - Efficacy of Steroids in Acute Vasogenic Edema
Brief Title: TBI- Efficacy of Steroids in Acute Vasogenic Edema
Acronym: TBI-SAVE
Status: Not yet recruiting | Type: Observational
Sponsor: Meditech Foundation (Other)
Responsible Party: Principal Investigator, Andres M. Rubiano, Medical and Research Director, Meditech Foundation
Other Study IDs: MF-2026-001; MF-2026-001 (Other Grant/Funding Number: Meditech Foundation)
Record Dates: First submitted 2026-01-02; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Traumatic Brain Injury
Keywords: Vasogenic Edema; Traumatic Brain Injury; Steroids; Brain Trauma
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Treatment Group: Patients with TBI and Dexamethasone Treatment after 5 days of Trauma
- Control Group: Patients with TBI without Dexamethasone Treatment after 5 days of Trauma

SUMMARY:
The goal of this observational study is to learn about the impact of dexamethasone treatment in traumatic brain injury patients with vasogenic edema in the second week after the trauma, administered in centers where this intervention has been considered to treat brain edema. The main question it aims to answer is: Does dexamethasone in a regimen of 8mg/8h for 5 days improve vasogenic edema in patients after 5 days of their trauma? Participants already receiving this treatment as part of their regular medical care in emergency settings, general wards, or ICU settings for TBI will be included, and data will be compared with patients with the same criteria but who do not receive the treatment.

DETAILED DESCRIPTION:
The present protocol proposes a Pragmatic Observational Treatment Clinical Trial (P-OCT) comparing the outcome of patients with TBI and brain contusions receiving dexamethasone in the vasogenic edema phase of TBI (days 5-6, at conventional doses of 8mg/8h for five days) and patients who traditionally do not receive steroids. The primary outcomes will include the Glasgow Outcome-Extended Score (GOSE) at discharge and one month after the event, including the evolution of clinical symptoms and findings obtained through non-invasive monitoring. This approach aims to generate evidence for a comprehensive physiopathology-based study, evaluating and already used medication with a new indication in a specific condition, that can be capable of modifying the management of vasogenic edema and subsequently the outcome of TBI patients.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70 years.
* Mild or moderate TBI, treated in the emergency department within the first 24-72 hours post-trauma.
* Abnormal CT scan with cerebral contusion, with or without midline shift >3 mm, and/or compression of basal cisterns.
* At least 2 systems with abnormal findings on non-invasive monitoring (ONSD ≥6 mm, reduced MCV, PI >1.3 or MCA FV <20cm/sec on transcranial Doppler, or ICP waveform with P2>P1).
* Patients with or without polytrauma, with an expected survival of>24 h.
* TBI with brain contusion with medical or surgical procedures indicated within the first 24 h (ventriculostomy, cisternostomy, decompressive craniectomy, or cranial decompression).

Exclusion Criteria:

* Age <18 or >70 years.
* Severe TBI (GCS = 3), suspected brain death, or head AIS = 6 (non-survivable injury).
* Normal CT scan on initial assessment.
* Clinical signs of cerebral herniation upon admission.
* Severe polytrauma or massive brain injury with an expected survival <24 h.
* Pre-existing neurological disorders that interfere with outcome assessment, preexisting conditions contraindicating steroid therapy or pre-existing conditions with permanent steroid therapy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include a prospective cohort of patients with TBI and no history of pre-existing neurological disorders that could interfere with outcome assessment. Patients must be treated in emergency departments within 24 to 72 hours after the traumatic event and need to have a CT scan ordered as part of the initial assessment. Patients must have a documented cerebral contusion on CT and evidence of progressive vasogenic edema confirmed by the initial and subsequent imaging. Patients can present clinical symptoms (headache, blurred vision, dizziness, nausea) and at least one documented abnormality in 2 non-invasive monitoring systems (ONSD ≥6 mm, pupillometry MCV reduced, transcranial Doppler with a PI >1.3 or an MCA flow velocity <20cm/sec, or ICP waveform with P2>P1 in any skull side)
Sampling Method: Probability Sample
Enrollment: 280 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2029-03-01 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
Score of every patient in the Glasgow Outcome Scale - Extended (GOS-E) one month after the event | 1 month after injury, assessed in person or by phone, according to the GOS-E manual (Wilson L et al. A Manual for the Glasgow Outcome Scale-Extended Interview. J Neurotrauma. 2021 Sep 1;38 (17):2435-2446. doi: 10.1089/neu.2020.7527. PMID: 33740873
  GOS-E Scoring system: Minimum Score = 1, Maximum Score = 8 Level 1 = Dead, Level 2 = Vegetative State:Condition of unawareness with only reflex responses, but with periods of spontaneous eye opening. Level 3 = Low Severe Disability; Level 4 = Upper Severe Disability: Patient who is dependent on daily support for mental or physical disability, usually a combination of both. If the patient can be left alone for more than 8 hours at home, it is the upper level of SD. If the patient cannot be left at home for more than 8 hours at home, it is a lower level of SD. Level 5 = Low Moderate Disability; Level 6 = Upper Moderate Disability: Patients have some disability such as aphasia, hemiparesis, or epilepsy and/or deficits of memory or personality, but can look after themselves. They are independent at home but dependent outside. If they can return to work even with special arrangements. GOS-E will be dichotomized into unfavorable outcome (GOS-E 1-6) and favorable outcome (GOS-E 7-8).

SECONDARY OUTCOMES:
Length of Stay in the Hospital | Since the time of the injury, up to 3 months
  Hospital Length of Stay, since the time of the injury, up to 3 months.

OTHER OUTCOMES:
Symptoms (blurred vision, headache, vomiting, dizziness, amnesia) | Since the injury, up to 3 weeks after the injury
  Type and number of symptoms after the treatment period, including blurred vision, headache, vomiting, dizziness, and amnesia. It will be taken from the medical records.
Infections (surgical site infection, pneumonia, urinary tract infections, meningitis, bacteremia) | Since the second week of the injury, up to 1 month after the injury
  Local or Systemic Infections, including surgical site infection, pneumonia, urinary tract infections, meningitis, and bacteremia. It will be recorded from the medical record.

CONTACTS AND LOCATIONS:
Overall Officials: Andres M Rubiano, MD, PhD, Principal Investigator — Meditech Foundation

IPD SHARING:
Plan to Share IPD: Yes
On Request
Supporting Information: Study Protocol, SAP, ICF
Time Frame: May 2029 - May 2034
Access Criteria: Researchers and Scientists, by request, to the officers' emails.
URL: http://www.meditechfoundationglobal.org

REFERENCES:
- [Background] Pérez-Bárcena J, Lara M, Pomar J, et al. DEXCON-TBI: protocol for a randomized controlled trial of dexamethasone in TBI. Trials. 2021;22(1):106
- [Background] Prasad GL, Pai A, Pt S. Short course of low-dose steroids for management of delayed pericontusional edema after mild traumatic brain injury - A retrospective study. Surg Neurol Int. 2025 Jan 24;16:23. doi: 10.25259/SNI_948_2024. eCollection 2025. PMID 39926471
- [Background] Moll A, Lara M, Pomar J, Orozco M, Frontera G, Llompart-Pou JA, Moratinos L, Gonzalez V, Ibanez J, Perez-Barcena J. Effects of dexamethasone in traumatic brain injury patients with pericontusional vasogenic edema: A prospective-observational DTI-MRI study. Medicine (Baltimore). 2020 Oct 23;99(43):e22879. doi: 10.1097/MD.0000000000022879. PMID 33120830
- [Background] Hutchinson PJ, Jalloh I, Helmy A, et al. The management of brain edema in traumatic brain injury: state of the art and future directions. Nat Rev Neurol. 2020;16(5):293-306
- [Background] Venkatesh B, Hickey RW, McDonald JR. Role of corticosteroids in acute brain injury revisited. Crit Care Med. 2020;48(11):1633-1642
- [Background] Edwards P, Arango M, Balica L, Cottingham R, El-Sayed H, Farrell B, Fernandes J, Gogichaisvili T, Golden N, Hartzenberg B, Husain M, Ulloa MI, Jerbi Z, Khamis H, Komolafe E, Laloe V, Lomas G, Ludwig S, Mazairac G, Munoz Sanchez Mde L, Nasi L, Olldashi F, Plunkett P, Roberts I, Sandercock P, Shakur H, Soler C, Stocker R, Svoboda P, Trenkler S, Venkataramana NK, Wasserberg J, Yates D, Yutthakasemsunt S; CRASH trial collaborators. Final results of MRC CRASH, a randomised placebo-controlled trial of intravenous corticosteroid in adults with head injury-outcomes at 6 months. Lancet. 2005 Jun 4-10;365(9475):1957-9. doi: 10.1016/S0140-6736(05)66552-X. PMID 15936423
- [Background] Cardona-Collazos S, Gonzalez WD, Pabon-Tsukamoto P, Gao GY, Younsi A, Paiva WS, Rubiano AM. Cerebral Edema in Traumatic Brain Injury. Biomedicines. 2025 Jul 15;13(7):1728. doi: 10.3390/biomedicines13071728. PMID 40722798
- [Background] Jha RM, Kochanek PM, Simard JM. Pathophysiology and treatment of cerebral edema in traumatic brain injury. Neuropharmacology. 2019 Feb;145(Pt B):230-246. doi: 10.1016/j.neuropharm.2018.08.004. Epub 2018 Aug 4. PMID 30086289